CLINICAL TRIAL: NCT00518128
Title: Measuring Effectiveness in Sleep Apnea Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Eric Kezirian, Associate Professor, Department of Otolaryngology--Head and Neck Surgery, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR024130
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Leptin; Homocysteine; C-reactive protein
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Surgical OSA Treatment Group: Moderate to Severe OSA patients who are unable to tolerate PAP (Positive Airway Pressure) and elect to proceed with surgical treatment (surgical cohort).
  Interventions: Procedure: Surgical OSA treatment
- 2 (Active Comparator): Positive Airway Pressure Therapy Comparison Group: Moderate to Severe OSA patients who tolerate PAP (Positive Airway Pressure).
  Interventions: Procedure: Positive Airway Pressure Therapy

INTERVENTIONS:
Procedure: Surgical OSA treatment — uvulopalatopharyngoplasty +/-tonsillectomy, genioglossus advancement, and hyoid suspension
  Other Names: UPPP, GA hyoid myotomy and suspension
  Arms: 1
Procedure: Positive Airway Pressure Therapy — Continuous positive airway pressure for treatment of obstructive sleep apnea
  Other Names: CPAP
  Arms: 2

SUMMARY:
The goal of this research is to improve our understanding of the effectiveness of surgical OSA treatment by evaluating its impact on these health-related and functional outcomes and comparing these effects to the changes in respiratory physiology achieved after surgery. To achieve this goal, we will examine key health-related (C-reactive protein, homocysteine, leptin, the homeostasis model of insulin resistance, and heart rate variability) and functional (sleep-related quality of life and vigilance) measures among a surgical group of OSA patients who do not tolerate non-surgical treatment (positive airway pressure, PAP) and a comparison group of matched OSA patients who tolerate PAP.

DETAILED DESCRIPTION:
The goal of this research is to improve our understanding of the effectiveness of surgical OSA treatment by evaluating its impact on these health-related and functional outcomes and comparing these effects to the changes in respiratory physiology achieved after surgery. To achieve this goal, we will examine key health-related (C-reactive protein, homocysteine, leptin, the homeostasis model of insulin resistance, and heart rate variability) and functional (sleep-related quality of life and vigilance) measures among a surgical group of OSA patients who do not tolerate non-surgical treatment (positive airway pressure, PAP) and a comparison group of matched OSA patients who tolerate PAP. We propose to measure the impact of surgical OSA treatment on these health-related and functional outcomes measures with the following three analyses: (1) to assess the changes seen with surgical treatment; (2) to compare changes seen with surgical and PAP treatment; and (3) to evaluate the association between changes in respiratory patterns during sleep and changes in health-related and functional outcomes measures for both surgical and PAP treatment.

ELIGIBILITY:
Inclusion Criteria (Surgical Group)

* Unable to tolerate PAP, supported by statement from sleep physician
* Multilevel airway obstruction
* Elect to proceed with surgical OSA treatment (uvulopalatopharyngoplasty +/-tonsillectomy, genioglossus advancement, and hyoid suspension)

Inclusion Criteria (Comparison Group-PAP)

* Tolerance of PAP during titration study and indication of willingness to use
* No previous treatment of PAP except during titration study
* Washout period of two weeks between PAP titration study and study assessment
* Matched to surgical group patient on age, gender, race, body mass index, and OSA disease severity (apnea-hypopnea index)

Exclusion Criteria:

* Pregnant women
* Primary snoring or mild OSA (apnea-hypopnea index < 15)
* Known neurologic, cardiac, hepatic, or renal disorder
* Acute illness or infection
* Co-existing sleep disorder other than primary snoring
* Unable to fast overnight prior to blood draw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
C-reactive protein level | Before and after surgery

SECONDARY OUTCOMES:
Leptin, Homocysteine, Homeostasis model of insulin resistance (HOMA-IR), Heart rate variability, Functional Outcomes of Sleep Questionnaire and Psychomotor Vigilance Task. | Before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kezirian, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Department of Otolaryngology - Head and Neck Surgery, San Francisco, California, United States

REFERENCES:
- [Derived] Kezirian EJ, Malhotra A, Goldberg AN, White DP. Changes in obstructive sleep apnea severity, biomarkers, and quality of life after multilevel surgery. Laryngoscope. 2010 Jul;120(7):1481-8. doi: 10.1002/lary.20946. PMID 20564750